CLINICAL TRIAL: NCT03518593
Title: Evaluation of NICHE (Nutritional Improvements Through Cash and Health Education) Programme Activities in Kitui and Machakos, Kenya
Brief Title: Evaluation of NICHE Programme Activities in Kenya
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kimetrica LLC (Industry)
Collaborators: UNICEF (Other); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UN-43203222
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Growth Disorders; Malnutrition
MeSH Terms: conditions — Growth Disorders; Malnutrition | interventions — CASP8 and FADD-Like Apoptosis Regulating Protein; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Additional cash transfer and nutritional counselling
  Interventions: Other: Cash and counselling
- Control (No Intervention): Existing cash transfer only

INTERVENTIONS:
Other: Cash and counselling — Additional 500 Ksh per child per month and household visits by Community health Volunteers (CHVs)
  Arms: Intervention

SUMMARY:
This study evaluates the impact of additional cash and nutritional counselling on nutrition outcomes in pregnant women and children up to the age of two years in CT-OVC (cash transfer- orphan and vulnerable children) households in Kitui and Machakos counties of Kenya. The control arm households will receive their normal CT-OVC cash payment and the intervention arm will receive an additional cash payment and nutritional counselling.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and children aged up to 23 months of age in households receiving CT-OVC cash transfers in Kitui and Machakos counties of Kenya

Exclusion Criteria:

* not residing in CT-OVC households

Max Age: 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-26 (Estimated); Study Completion 2018-06-26 (Estimated)

PRIMARY OUTCOMES:
Stunting | 8-15 months
  HAZ (height for age z score) < -2 SDs of WHO median

CONTACTS AND LOCATIONS:
Overall Officials: Helen Guyatt, PhD, Principal Investigator — Kimetrica LLC

IPD SHARING:
Plan to Share IPD: Undecided